CLINICAL TRIAL: NCT04046354
Title: Clinical Trial of Microwave Ablation System
Brief Title: Microwave vs. Radiofrequency Ablation for Benign Thyroid Nodules: A Multicenter Randomized Controlled Trial Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu Jie, Associate chief physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2018001
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Benign Thyroid Nodules; Ablation
Keywords: microwave; thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The group will use microwave ablation equipment to treat benign thyroid nodules.
  Interventions: Device: Ultrasound-guided Percutaneous Microwave Ablation
- Group B (Active Comparator): The group will use radiofrequency ablation equipment to treat benign thyroid nodules.
  Interventions: Device: Ultrasound-guided Percutaneous Radiofrequency Ablation

INTERVENTIONS:
Device: Ultrasound-guided Percutaneous Microwave Ablation — Ultrasound-guided Percutaneous Microwave Ablation
  Arms: Group A
Device: Ultrasound-guided Percutaneous Radiofrequency Ablation — Ultrasound-guided Percutaneous Radiofrequency Ablation
  Arms: Group B

SUMMARY:
Compared with traditional treatment methods, ultrasound-guided thermal ablation is more targeted, less invasive and more reliable. The study compared microwave ablation and radiofrequency ablation to evaluate the efficacy and safety in the treatment of benign thyroid nodules with a multicenter data, which will provide a basis for clinical treatment.

DETAILED DESCRIPTION:
Ultrasound-guided minimally invasive treatment has accurate positioning, higher targeting, no need for general anesthesia, less trauma for patients, and more reliable efficacy.Currently, it mainly includes percutaneous anhydrous ethanol injection, radiofrequency ablation and microwave ablation for the treatment of thyroid nodules.Currently, radiofrequency ablation and microwave ablation are mainly used to treat thyroid nodules.

This study was a randomized, parallel, positive control, and non-inferiority multicenter clinical study.Radiofrequency ablation was used as the positive control.Follow-up was conducted at 1, 3, 6 and 12 months after ablation. The primary endpoint was the rate of nodule volume reduction at 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years and ≤75 years
* The pathological diagnosis was benign thyroid nodules within 6 months
* Diameter ≥2cm, solid > 80%, the number of multiple nodules≤ 3
* Participate voluntarily and sign the informed consent

Exclusion Criteria:

* Coagulation mechanism disorder or bleeding tendency
* Patients with severe cardiopulmonary insufficiency
* Blood pressure cannot be effectively controlled
* abnormal liver function
* Blood glucose cannot be effectively controlled
* Abnormal thyroid function
* Allergic history of ultrasound contrast agent
* Suspicious lymph node metastasis in the cervical region
* Abnormal contralateral vocal cord function
* Pregnant and lactating women
* Have participated in clinical trials of any drug and/or medical device within 3 months prior to enrollment
* The researchers believe that there are any other factors that are not suitable for inclusion or that affect participants' participation in the study.
* Patients with inner pacemaker, hearing aid, metal stent, titanium clip, internal (external) steel plate and other metal objects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume reduction rate of thyroid nodules | up to 12 months.
  volume reduction rate，VRR=(Volume before treatment - volume at follow-up)/Volume before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yu, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rastogi A, Bhadada SK, Bhansali A. Nodular goiter with multiple cystic and solid swellings. Indian J Endocrinol Metab. 2012 Jul;16(4):651-3. doi: 10.4103/2230-8210.98034. PMID 22837936
- [Background] Kihara M, Hirokawa M, Masuoka H, Yabuta T, Shindo H, Higashiyama T, Fukushima M, Yamada O, Takamura Y, Ito Y, Kobayashi K, Miya A, Miyauchi A. Evaluation of cytologically benign solitary thyroid nodules by ultrasonography: a retrospective analysis of 1877 cases. Auris Nasus Larynx. 2013 Jun;40(3):308-11. doi: 10.1016/j.anl.2012.09.007. Epub 2012 Oct 24. PMID 23103151
- [Background] Wright AS, Sampson LA, Warner TF, Mahvi DM, Lee FT Jr. Radiofrequency versus microwave ablation in a hepatic porcine model. Radiology. 2005 Jul;236(1):132-9. doi: 10.1148/radiol.2361031249. PMID 15987969
- [Derived] Chen S, Dou J, Cang Y, Che Y, Dong G, Zhang C, Xu D, Long Q, Yu J, Liang P. Microwave versus Radiofrequency Ablation in Treating Predominantly Solid Benign Thyroid Nodules: A Randomized Controlled Trial. Radiology. 2024 Oct;313(1):e232162. doi: 10.1148/radiol.232162. PMID 39436295